CLINICAL TRIAL: NCT00675233
Title: Phase I Trial of Photodynamic Therapy With HPPH (2-1[Hexyloxyethyl]-2-devinylpyropheophorbide-a) for Treatment of Dysplasia, Carcinoma in Situ and T1 Carcinoma of the Larynx
Brief Title: Photodynamic Therapy Using HPPH in Treating Patients With Dysplasia, Cancer in Situ, or Invasive Cancer of the Larynx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595166; I 119207
Record Dates: First submitted 2008-05-08; First posted 2008-05-09 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage 0 laryngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment PDT (Experimental): Patients undergo PDT comprising HPPH IV over 1 hour on day 1 followed by laser light to the tumor on day 2. At least 6 weeks later, patients achieving partial response, no response, or a geographical miss may undergo a second course of treatment.
  Interventions: Drug: HPPH; Procedure: laser therapy

INTERVENTIONS:
Drug: HPPH — Given IV
Procedure: laser therapy — Escalating light doses with 665 nm light

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as HPPH, that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. This may be an effective treatment for laryngeal cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of laser light therapy when given together with HPPH in treating patients with dysplasia, cancer in situ, or invasive cancer of the larynx.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of laser light therapy using a fixed dose of HPPH in patients with dysplasia, squamous cell carcinoma in situ, or T1 squamous cell carcinoma of the larynx.

Secondary

* To determine response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of laser light therapy.

Patients undergo photodynamic therapy comprising HPPH IV over 1 hour on day 1 and laser light therapy to the tumor on day 2. Approximately 8 weeks later, patients with a partial response, no response, or a geographical miss may receive a second course of treatment.

After completion of study treatment, patients are followed at 1 week, 1 month, 3 months, and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-confirmed diagnosis of 1 of the following:

  * Mild to severe dysplasia of the larynx

    * Dysplastic lesions > 3 mm in thickness
  * Squamous cell carcinoma in situ of the larynx
  * T1 squamous cell carcinoma of the larynx

    * Tumor > 3 mm in thickness
    * No T2-T4 squamous cell carcinoma of the larynx
* Newly diagnosed or recurrent disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin > 2.0 mg/dL
* Creatinine > 2.0 mg/dL
* SGOT > 3 times upper limit of normal (ULN)
* Alkaline phosphatase > 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3-6 months after completion of study treatment
* No porphyria
* No hypersensitivity to porphyrin or porphyrin-like compounds

PRIOR CONCURRENT THERAPY:

* Any prior therapy allowed
* At least 4 weeks since prior and no concurrent chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-04-25 (Actual); Primary Completion 2013-06-28 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Toxicity | 6 weeks
Tumor response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States